CLINICAL TRIAL: NCT01227122
Title: Plasmatic Level of Neutrophil Gelatinase-Associated Lipocalin (NGAL) as a Predictive Marker of Acute Kidney Failure in Patients With Preoperative Chronic Kidney Failure Undergoing Cardiac Surgery.
Brief Title: NGAL Predictive Value of Acute Kidney Failure After Cardiac Surgery in Patients With Preoperative Chronic Kidney Failure
Acronym: NGAL-CKF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hopital Jean Minjoz (Other)
Responsible Party: Principal Investigator, Prof. Sidney Chocron, MD, PhD, Hopital Jean Minjoz
Other Study IDs: 2010-A00111-38
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Preoperative KIDNEY FAILURE, CHRONIC; Postoperative KIDNEY FAILURE, ACUTE; Cardiac Surgical Procedures
Keywords: NGAL plasmatic level; Preoperative KIDNEY FAILURE, CHRONIC; Postoperative KIDNEY FAILURE, ACUTE; Cardiac Surgery Procedures
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Primary endpoint: To evaluate predictive value of plasmatic levels of Neutrophil Gelatinase Associated Lipocalin (NGAL) to reveal acute kidney failure after cardiac surgery in patients with preoperative chronic kidney failure Secondary endpoint is to obtain threshold values of NGAL.

DETAILED DESCRIPTION:
(N/A)

ELIGIBILITY:
Inclusion Criteria:

* Renal clearance less than 60 mL/min
* Able to give written consent
* Elective valve surgery
* Elective CABG surgery

Exclusion Criteria:

* Less than 18 years old
* Iodine injection within 3 days before surgery
* Iodine injection within 24 first postoperative hours
* preoperative infection
* evolutive cancer disease
* Refusal
* Pregnancy
* Unable to give written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a chronic kidney failure, undergoing cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-08; Primary Completion 2013-07 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Neutrophil Gelatinase Associated Lipocalin (NGAL) level | From surgery to discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Chocron Sidney, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire (CHU) Jean Minjoz, Besançon, France
Locations (1):
- Centre hospitalier Universitaire (CHU) Jean Minjoz, Besançon, Franche-Comté, France